CLINICAL TRIAL: NCT02734199
Title: Highly Effective Reversible Contraceptive Initiative-Salt Lake (HER-SL)
Brief Title: HER Salt Lake Initiative
Acronym: HER-SL
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: William and Flora Hewlett Foundation (Other); Society of Family Planning (Other)
Responsible Party: Principal Investigator, David Turok, Principal Investigator, University of Utah
Other Study IDs: 67378
Record Dates: First submitted 2016-03-08; First posted 2016-04-12 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Birth Control; Contraception
Keywords: Birth Control; Contraception; IUD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Enrollment Period 1 Cohort: Cohort 1 includes approximately 650 participants who receive a standardized client centered contraceptive counseling session with a clinical assistant. Contraceptive access will be the same as it was prior to the study beginning, meaning participants either have to use insurance or self-pay for their method of choice.
- Enrollment Period 2 Cohort: Cohort 2 includes approximately 1000 participants who receive a standardized client centered contraceptive counseling session with a clinical assistant. Financial barriers are removed for Period 2 participants and they can initiate which ever contraceptive method they want at no cost to them for three years.
- Enrollment Period 3 Cohort: Cohort 3 includes approximately 1350 participants who receive a standardized client centered contraceptive counseling session with a clinical assistant. Financial barriers are removed for Period 3 participants and they can initiate which ever contraceptive method they want at no cost to them for three years. During enrollment period 3, a community-wide, media driven intervention will be implemented and population level changes in HER-C initiation will be examined.

SUMMARY:
This study aims to understand the long-term health, social, and economic impacts of transitioning a community to Highly Effective Reversible Contraception (HER-C).

DETAILED DESCRIPTION:
The persistently high rate of unintended pregnancy in the US suggests an inadequacy of current prevention models and a need for new approaches to contraceptive acceptability and promotion. Although popularity of Highly Effective Reversible Contraception (HER-C) in the US is steadily increasing, less than 10% of contracepting women use intrauterine devices (IUDs) or subdermal contraceptive implants, which are the most effective methods for avoiding unintended pregnancy.

Poverty is an important predictor of unintended pregnancy where women with incomes below the Federal Poverty Level (FPL) have over a five-fold increased risk of unintended pregnancy relative to women with higher incomes. Because of limited public funds for family planning, low-income women in Salt Lake County have limited access to HER-C, which has high initiation cost but significant cost-saving potential over time. Additionally, contraceptive research has inadequately measured the social impact of HER-C.

The first aim of the HER Salt Lake Initiative is to evaluate the increase in HER-C methods with three strategies: 1) Client centered contraceptive counseling; 2) Removal of financial barriers; and 3) Targeted media campaigns.

The second aim of the HER Salt Lake Initiative is to assess changes in earnings and education among women initiating HER-C compared to other methods of contraception and model the projected lifetime earning potential of women based on their contraceptive method choices.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 16-45 years of age
* Seeking contraceptive counseling and services at four participating Planned Parenthood clinics in Salt Lake County
* Desire to prevent pregnancy for at least one year
* Fluent in English or Spanish
* Their current preferred phone number must be functioning at the time of study entry and will be tested prior to enrollment

Exclusion Criteria:

* Currently pregnant and planning to continue the pregnancy, or trying to get pregnant
* Relying on female or male sterilization as contraceptive method

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Females 16-45 years of age, who desire to prevent pregnancy for at least one year and are seeking contraceptive counseling and long term contraception services in Salt Lake County.
Sampling Method: Non-Probability Sample
Enrollment: 4430 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Contraceptive method choice and continuation per participant report and medical record documentation | at enrollment through 36 months
  Assess contraceptive method choice and use in relation to participant demographic and socioeconomic characteristics at enrollment, 12 months, 24 months, and 36 months.

SECONDARY OUTCOMES:
Federal Poverty Level (FPL) status by participant reported income | at enrollment through 36 months
  Assess Federal Poverty Level (FPL) at enrollment and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: David K Turok, MD, Principal Investigator — University of Utah, Department of Obstetrics & Gynecology
Locations (1):
- Planned Parenthood Association of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simmons RG, Carter G, Sanders JN, Turok DK. Assessing Contraceptive Switching and Discontinuation Over 3 Years in the HER Salt Lake Study. Obstet Gynecol. 2024 Jul 1;144(1):79-88. doi: 10.1097/AOG.0000000000005621. Epub 2024 May 23. PMID 38781634
- [Derived] Gero A, Simmons RG, Sanders JN, Turok DK. Does access to no-cost contraception change method selection among individuals who report difficulty paying for health-related care? BMC Womens Health. 2022 Aug 2;22(1):327. doi: 10.1186/s12905-022-01911-x. PMID 35918666
- [Derived] Higgins JA, Kramer R, Senderowicz L, Everett B, Turok DK, Sanders JN. Sex, poverty, and public health: Connections between sexual wellbeing and economic resources among US reproductive health clients. Perspect Sex Reprod Health. 2022 Mar;54(1):25-28. doi: 10.1363/psrh.12189. Epub 2022 Feb 27. PMID 35220665
- [Derived] Dalessandro C, Kaiser J, Sanders JN. Reproductive autonomy and feelings of control over pregnancy among emerging adult clients in a Utah (USA) contraceptive initiative study. Sex Reprod Healthc. 2022 Mar;31:100688. doi: 10.1016/j.srhc.2021.100688. Epub 2021 Nov 26. PMID 34864316
- [Derived] Kramer RD, Higgins JA, Everett B, Turok DK, Sanders JN. A prospective analysis of the relationship between sexual acceptability and contraceptive satisfaction over time. Am J Obstet Gynecol. 2022 Mar;226(3):396.e1-396.e11. doi: 10.1016/j.ajog.2021.10.008. Epub 2021 Oct 14. PMID 34656551
- [Derived] Myers K, Sanders JN, Dalessandro C, Sexsmith CD, Geist C, Turok DK. The HER Salt Lake media campaign: comparing characteristics and outcomes of clients who make appointments online versus standard scheduling. BMC Womens Health. 2021 Mar 23;21(1):121. doi: 10.1186/s12905-021-01256-x. PMID 33757511
- [Derived] Simmons RG, Sanders JN, Geist C, Gawron L, Myers K, Turok DK. Predictors of contraceptive switching and discontinuation within the first 6 months of use among Highly Effective Reversible Contraceptive Initiative Salt Lake study participants. Am J Obstet Gynecol. 2019 Apr;220(4):376.e1-376.e12. doi: 10.1016/j.ajog.2018.12.022. Epub 2018 Dec 18. PMID 30576664
- [Derived] Higgins JA, Sanders JN, Palta M, Turok DK. Women's Sexual Function, Satisfaction, and Perceptions After Starting Long-Acting Reversible Contraceptives. Obstet Gynecol. 2016 Nov;128(5):1143-1151. doi: 10.1097/AOG.0000000000001655. PMID 27741195